CLINICAL TRIAL: NCT04593589
Title: Autologous Transplantation of Adult Salivary Gland Stem Cells to Restore Submandibular Gland Function After Radiotherapy
Brief Title: Submandibular Gland Stem Cell Transplantation
Acronym: RESTART
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RT2020-04; NL75095.000.20 (Registry Identifier: CCMO register)
Record Dates: First submitted 2020-09-04; First posted 2020-10-20 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-09

CONDITIONS: Head and Neck Cancer
Keywords: Radiotherapy; Cell transplantation; Stem cell therapy
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Transplantation (Experimental): Submandibular Gland Stem Cell Transplantation
  Interventions: Other: Submandibular Gland Stem Cell Transplantation

INTERVENTIONS:
Other: Submandibular Gland Stem Cell Transplantation — Autologous transplantation of salivary stem cells (salisphere derived cells) cultured in vitro as obtained from submandibular glands after postoperative radiotherapy

SUMMARY:
This study is a phase I safety and feasibility study to treat head and neck cancer patients with autologous salivary gland stem cell transplantation after postoperative (chemo)radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Squamous cell carcinoma (SCC) originating from the mucosa of the oral cavity;
* Primary resection of tumour including an electively or therapeutic ipsilateral neck dissection (at least levels Ib to III, including the submandibular gland).
* Postoperative radiotherapy or chemoradiation, including prophylactic or therapeutic irradiation of the contralateral side of the neck (where the remaining submandibular gland is), including at least levels Ib to IV), next to irradiation of the tumour bed and ipsilateral neck (current standard);
* Age ≥ 18 years;
* WHO performance 0-2;
* Written informed consent;

Exclusion Criteria:

* Primary (definitive) radiotherapy, with or without systemic treatment;
* Previous radiotherapy of the head and neck region (re-irradiation);
* Positive microbiological screening for Human Immunodeficiency Virus type 1 and 2, hepatitis B and C virus and Treponema pallidum.
* Presence of systemic disease known to affect salivary gland functioning (e.g., Sjögren's syndrome);
* Known allergy to mice and gentamicin
* History within the past five years of malignancies other than:

  * basal or squamous cell carcinoma of the skin
  * in situ carcinoma of the cervix;
* Females who are pregnant or lactating at entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-05-10 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Safety: adverse events | Data for assessing safety will be recorded from day 1 to 365.
  The number of adverse events (AE), serious adverse events (SAE) or suspected unexpected adverse reactions (SUSAR) after autologous salivary stem cell transplantation. All possible adverse events will be scored according to the definitions of the Common Toxicity Criteria for Adverse Events version 4.0 (CTCAEv4.0).
Feasibility: salivary flow rate | Data for assessing feasibility will be recorded 6 and 12 months after autologous stem cell transplantation to assess if salivary flow will be increased compared to salivary flow before transplantation.
  The salivary flow rate of the remaining submandibular gland will be recorded.

SECONDARY OUTCOMES:
Salivary flow recovery | Saliva measurements at 6 and 12 months and then on a yearly basis until 5 years after postoperative (chemo)radiation
  Unstimulated whole saliva, paraffin stimulated whole saliva and 5% citric acid stimulated parotid and submandibular/sublingual saliva measurements.
Impact of transplantation | Patient-rated outcome measures at 6 and 12 months and then on a yearly basis until 5 years after postoperative (chemo)radiation
  Patient-rated outcome measures including various side effects related to the postoperative (chemo)radiation and Quality of Life (QoL) using internationally validated questionnaires.
Locoregional control | 5 years after postoperative (chemo)radiation
  Locoregional control is defined as the number of patients with recurrent disease within or adjacent to the primary tumor site and regional lymph nodes after postoperative (chemo)radiation, assessed by pathology and/or oncologic imaging (CT, MRI or PET).
Overall survival and disease-free survival | 5 years after postoperative (chemo)radiation
Rate of water diffusion in remaining submandibular gland | 6 and 12 months after postoperative (chemo)radiation
  The rate of water diffusion in remaining submandibular gland derived from DWI/DTI-MRI.
Amount of PSMA | 6 and 12 months after autologous stem cell transplantation
  The amount of prostate specific membrane antigen (PSMA) in the remaining submandibular gland derived from PET-CT

CONTACTS AND LOCATIONS:
Overall Officials: R.J.H.M. Steenbakkers, MD, PhD, Principal Investigator — UMC Groningen
Locations (1):
- UMCG, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No